CLINICAL TRIAL: NCT01131377
Title: Acetazolamide Facilitates Ventilator Weaning Multicenter, Prospective, Double Blinded, Randomised Controlled Trial
Brief Title: Acetazolamide Facilitates Ventilator Weaning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Chae-Man Lim/Department of Pulmonary and Critical Care Medicine, Asan Medical Center, University of Ulsan College of Medicine, Seoul, Korea, Department of Pulmonary and Critical Care Medicine, Asan Medical Center, University of Ulsan College of Medicine, Seoul, Korea
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AMCAZM-150
Record Dates: First submitted 2010-05-26; First posted 2010-05-27 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2010-04

CONDITIONS: Ventilator Weaning; Alkalosis, Metabolic
Keywords: mechanical ventilation weaning phase patients with metabolic alkalosis
MeSH Terms: conditions — Alkalosis | interventions — Acetazolamide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acetazolamide (Experimental): If ABGA is pH ≥ 7.43 & HCO3- ≥ 26mEq/L at 7am, they will receive acetazolamide 500mg via IV.
  If ABGA is pH ≤ 7.35 at 7am, acetazolamide will skip.
  Interventions: Drug: acetazolamide
- Placebo (Placebo Comparator): This group will be managed with general metabolic alkalosis treatment such as electrolyte correction, hydration except acetazolamide.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: acetazolamide — If ABGA is pH ≥ 7.43 & HCO3- ≥ 26mEq/L at 7am, they will receive acetazolamide 500mg via IV q 24h.
  If ABGA is pH ≤ 7.35 at 7am, acetazolamide will skip.
  Other Names: acetazolamide = Zoladin
  Arms: Acetazolamide
Drug: Saline — They will receive saline 50ml via IV q 24h.
  Arms: Placebo

SUMMARY:
Metabolic alkalosis(MA) is common metabolic disorder in ICU setting. MA could be cause of weaning failure or delay by depression of respiratory center. The purpose of this study is to evaluate that correction of MA by administration of acetazolamide facilitates weaning of mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Patients on mechanical ventilation for at least 24 hours with an assisted mode and passed acute resuscitation and considered for weaning. (Definition of Weaning point:

  1. Oxygenation

     * FiO2 ≤ 0.4 & PaO2 ≥ 60 mmHg

       * O2 index (PaO2/FiO2) ≥ 150

         * SaO2 > 90%

           * PEEP ≤ 5 cmH2O

             * MN ≤ 15 L/min
  2. Vital sign

     * Stable BP: MAP ≥ 60 mmHg ((i.e., no epinephrine or norepinephrine <0.2μg/kg/min, or equivalent dose vasopressin or phenylephrine)

       * HR ≤ 140bpm

         * 35 ≤ BT ≤ 38 ℃

           * RR ≤ 35/min
  3. Clinical status

     * resolution of acute disease process

       * no newly developed pulmonary infiltration

         * Ramsay sedation score 2~4

           * Hb > 7, pH > 7.30, normal electrolyte

             * no active bleeding, no IICP, no bronchospasm, no CAD

               * no rescure or specific treatment (NO, prone, OP plan)
* ABGA : pH ≥ 7.43 and HCO3- ≥ 26mEq/L

Exclusion Criteria:

* Permanent ventilator dependency due to brainstem disease, diffuse cerebral disease, severe respiratory or neuromuscular disease
* Active bleeding, IICP, unstable coronary artery disease, bronchospasm, and rescue treatment (inhaled NO, prone), pre-op condition
* Contraindication to acetazolamide: renal insufficiency (creatinine clearance <20 ml/min and/or renal replacement therapy), intolerance or allergy to acetazolamide or sulfonamides, hyperchloremic metabolic acidosis, hyponatremia (Na<130), hypokalemia (K<3.5), adrenal insufficiency.
* Diaphragm dysfunction : as diagnosed by fluoroscopy, nerve conduction velocity, USG, or overt paradoxical motion of the abdomen

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-05 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
weaning time between two group | hour
  Weaning time : [total ventilation time] - [total controlled mode time]

SECONDARY OUTCOMES:
Successful weaning rate between two group
  Successful weaning : self respiration more than 48h after withdrawl mechanical ventilation
total duration of mechanical ventilation between two group | hour
length of ICU stay between two group | hour
frequency of ventilator associated pneumonia between two group
overall ICU mortality between two group

CONTACTS AND LOCATIONS:
Overall Officials: Chae-Man Lim, professor, Study Chair — Department of Pulmonary and Critical Care Medicine, Asan Medical Center, University of Ulsan College of Medicine, Seoul, Korea
Locations (1):
- AMC MICU; Asan medical center, Seoul, 388-1, Pungnap-dong, Songpa-gu, South Korea